CLINICAL TRIAL: NCT00004985
Title: A Phase II, Single-Blind, Randomized, Placebo-Controlled Study of Capravirine (AG1549) in Combination With Viracept and Two Nucleoside Reverse Transcriptase Inhibitors in HIV-Infected Subjects Who Failed an Initial Nonnucleoside Reverse Transcriptase Inhibitor Containing Regimen
Brief Title: Combination Treatment Using Capravirine (AG1549), Nelfinavir, and Two Nucleoside Reverse Transcriptase Inhibitors in HIV Patients Who Failed Initial Combination Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Agouron Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 286D; AG1549-509
Record Dates: First submitted 2000-03-15; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-03

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; HIV Protease Inhibitors; RNA, Viral; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; Nelfinavir
MeSH Terms: conditions — HIV Infections | interventions — capravirine; Nelfinavir

INTERVENTIONS:
Drug: Capravirine
Drug: Nelfinavir mesylate

SUMMARY:
The purpose of this study is to look at the effectiveness of an anti-HIV drug combination that adds capravirine in patients who have failed their first drug combination treatment.

DETAILED DESCRIPTION:
[Note: As of 2/28/2001, due to toxicity studies and concern for safety, changes in the methodology were implemented and patients need to sign new informed consents. The study is unblinded. Group 1 receives AG1549; Group 2 receives an AG1549 placebo. Patients who are taking capravirine and who currently have viral loads below 400 copies/ml may continue to take capravirine at 1400 mg twice daily. Capravirine will be discontinued in patients with viral loads greater than 400 copies/ml at their last visit and they will be switched to new therapies or continue with their background therapies as deemed appropriate by the investigators.] Both groups also receive nelfinavir mesylate and 2 NRTIs. All patients receive the same dose of nelfinavir mesylate. The NRTIs are selected at the investigator's discretion provided the patient has not previously received the chosen NRTIs. Patients have regular physical examinations. Blood samples are collected regularly and at 1 month post-treatment to determine plasma HIV RNA, pharmacokinetics, and CD4 and CD8 counts. Patients who complete 24 weeks of treatment will have the option to continue treatment for an additional 24 weeks or end participation.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this trial if they:

* Are HIV-positive.
* Have a CD4 cell count more than 50/mm3.
* Are at least 18 years old.
* Have adequate blood, kidney, and liver functions.
* Are currently taking an anti-HIV drug combination of an NNRTI plus 1 or more NRTIs for more than 28 days and are failing that combination.

Exclusion Criteria

Patients will not be eligible for this trial if they:

* Have had any protease inhibitor or capravirine treatment.
* Have been given any drug that interferes with their immune system or with the study drugs within 28 days of study entry.
* Have had radiation therapy within 28 days of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75
Dates: Start 2000-01

CONTACTS AND LOCATIONS:
Locations (34):
- United States (33):
  - Phoenix Body Positive, Phoenix, Arizona
  - Pacific Oaks Med Group, Beverly Hills, California
  - First Choice Medical, Palm Springs, California
  - Apogee Med Group, San Diego, California
  - Saint Francis Mem Hosp / HIV Care Unit, San Francisco, California
  - Kaiser Foundation Hospital, San Francisco, California
  - Harbor - UCLA Med Ctr, Torrance, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Bach and Godofsky, Bradenton, Florida
  - Clin Research of West Florida, Clearwater, Florida
  - Community Health Care, Fort Lauderdale, Florida
  - Therafirst Med Ctr, Fort Lauderdale, Florida
  - South Shore Hosp, Miami, Florida
  - Immunity Care and Research Inc, Miami Beach, Florida
  - Orange County Health Dept, Orlando, Florida
  - Infectious Diseases Associates, Sarasota, Florida
  - Hillsborough County Health Dept, Tampa, Florida
  - Treasure Coast Infectious Disease Consultants, Vero Beach, Florida
  - Polk County Health Dept, Winter Haven, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Braude Mermin Spivey MD PC, Atlanta, Georgia
  - Massachusetts Gen Hosp, Boston, Massachusetts
  - Fenway Community Health Ctr, Boston, Massachusetts
  - VAMC New Jersey Healthcare System, East Orange, New Jersey
  - Jersey Shore Med Ctr, Neptune City, New Jersey
  - Infectious Disease Assoc of Central Jersey, Somerville, New Jersey
  - Biomedical Research Alliance of New York, Jamaica, New York
  - North Shore Univ Hosp, Manhasset, New York
  - Liberty Medical, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Central Texas Clinical Research, Austin, Texas
  - Univ TX Galveston Med Branch, Galveston, Texas
  - Infectious Disease Physicians Inc, Annandale, Virginia
- Clinical Research Puerto Rico Inc, San Juan, Puerto Rico